CLINICAL TRIAL: NCT03302468
Title: Development and Validation of the Endometriosis Health Profile-30 Traditional Chinese (Hong Kong) Version in Endometriosis and Adenomyosis
Brief Title: Development and Validation of EHP-30 (Hong Kong Chinese Version) for Patients With Endometriosis and Adenomyosis
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fung Wen Ying Linda, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: EHP30 traditional Chinese
Record Dates: First submitted 2017-09-18; First posted 2017-10-05 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis; Adenomyosis
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Endometriosis and adenomyosis can impact on the quality of life including the physical, psychological and social aspects. It is important to include quality of life measurements in evaluating the disease severity and response to any given treatment. The 30-item Endometriosis Health Profile (EHP-30), derived from in-depth interviews of patients with endometriosis, is currently the most reliable questionnaire for health-related quality of life measurement in women with endometriosis. It includes specific questions addressing the problems faced by patients with endometriosis.

Unfortunately, this widely accepted tool does not have a traditional Chinese version for the measurement of health-related quality of life of endometriosis in Hong Kong. Furthermore, adenomyosis and endometriosis share similar histological and clinical symptomatology, but application of EHP-30 to adenomyosis has never been studied.

The aims of the present study are to translate the EHP-30 English version into traditional Chinese version and to evaluate its psychometric properties in endometriosis and adenomyosis.

The hypothesis of this study is that EHP-30 (Hong Kong) traditional Chinese questionnaire has high internal consistency, construct validity, reproducibility as the original English version and can be applicable to Hong Kong Chinese women with endometriosis and adenomyosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic condition caused by the presence of ectopic endometrial tissue outside the uterus, affecting the fallopian tubes, ovaries, pelvic peritoneum or even the urinary and gastrointestinal tracts. Adenomyosis is characterized by the presence of ectopic endometrial gland and stroma in the myometrium with associated myometrial hypertrophy and hyperplasia. Adenomyosis has been reported to occur in 30-60% of the hysterectomy specimen.Endometriosis causes painful symptoms including dysmenorrhoea, pelvic pain, dyspareunia and infertility. Adenomyosis also causes clinically significant symptoms include dysmenorrhoea, pelvic pain and heavy menstrual flow.

Both conditions can impact on the quality of life including the physical, psychological and social aspects. It is important to include quality of life measurements in evaluating the disease severity and response to any given treatment. The 30-item Endometriosis Health Profile (EHP-30), derived from in-depth interviews of patients with endometriosis, is currently the most reliable questionnaire for health-related quality of life measurement in women with endometriosis. It includes specific questions addressing the problems faced by patients with endometriosis. It also exhibits good reliability, validity and interpretability.

The EHP-30 has recently been translated into simplified Chinese version and evaluated with psychometric tests which showed the simplified Chinese version is a valid, reliable and acceptable tool for the measurement of the health-related quality of life of women with endometriosis in mainland China. Unfortunately, this widely accepted tool does not have a traditional Chinese version for the measurement of health-related quality of life of endometriosis in Hong Kong. Furthermore, adenomyosis and endometriosis share similar histological and clinical symptomatology, but application of EHP-30 to adenomyosis has not been studied. The aims of the present study are to translate the EHP-30 English version into traditional Chinese version and to evaluate its psychometric properties in endometriosis and adenomyosis.

EHP-30 consists of 30 items in English, grouping into five subscales measuring pain (11 items), control and powerlessness (6 items), emotions (6 items), social support (4 items) and self-image (3 items) in part one. Part two consists of 23 items, grouping into six subscales may not be applicable to all adenomyosis patients: work (5 items), relationship with children (2 items), sexual intercourse (5 items), medical profession (4 items), treatment (3 items) and infertility (4 items). Participants choose their response from a five point likert scale from 0 to 4. Items within each subscale will be added up to generate a subscale score. Then, the subscale score is divided by maximum possible score and multiply by 100 to give a health status score which 100 represent worst health and 0 represent best health status.

Firstly, approval to use EHP-30 will be obtained from the original author, Dr Georgina Jones. We will adhere to the Good Practice for the Translation and Cultural adaptation process for patient-reported outcomes measures guideline. 6 The EHP-30 will be evaluated by 2 bilingual researchers in the fields of gynaecology independently and decide if any item will be regarded as inappropriate. They will then perform the forward translation of the EHP-30 to traditional Chinese independently. After that, they will review the two versions of translation and hold a meeting for discussion on items of discrepancy, in order to produce one version. Back-translation will be performed by another 2 persons who are professional in Chinese-English translation, after the iterative evaluation of forward translation process. The original and back-translated versions will be compared for accuracy and comprehension by another two monolingual researchers. If substantial differences existed between the two original and the back-translated versions, the translation-back translation process are repeated until a questionnaire representative of the original is obtained. Finally, the back-translated version will be sent to Dr Georgina Jones and the colleagues. Comments on the back-translated version will be obtained from them.

Pilot phase of the translated questionnaire Chinese women attending the Gynaecology clinic of New Territories East Cluster with pelvic painful symptoms will be invited to join the study. Exclusion criteria include an age of less than 18 years, mental incapacity that would preclude completion of the questionnaire and those who refuse to join. Written consent will be obtained from them by a research assistant. They will be asked to complete the EHP-30 and SF-36 at the specialty clinic. After filling in the questionnaires, they will be asked to give comments on the questionnaire.

Any patient attending the gynaecology clinic who fulfills the inclusion criteria and without any exclusion criteria will be invited for participation in the study. If the patient is willing to participate, written consent will be obtained from the patient. The study investigators will record demographic features and characteristics of the disease. The patient will be asked to complete the traditional-Chinese version of EHP-30 and traditional-Chinese version of the Medical Outcomes Study Short Form 36-item health survey (SF-36). 11-13 Demographic data collected include age, height, weight, education level, marital status, monthly household income and employment status. Disease characteristics for endometriosis include intensity of painful symptoms by visual analog scale (VAS), menstrual blood loss by pictorial blood loss assessment chart (PBAC) and intraoperative scoring of the severity of endometriosis. Disease characteristics for adenomyosis include VAS scores on painful symptoms, size of uterus and size of adenomyosis and menstrual blood loss by pictorial blood loss assessment chart (PBAC).

Exploring the impact of quality of life is important to clinical practice. The Medical Outcomes Study Short Form 36-item health survey (SF-36) is a generic type of Health Related Quality of Life (HRQoL) assessment tool widely used in different disease conditions. Questionnaire which assesses eight dimensions of QoL of an individual. A higher score means a better quality of life. It has been used to study QoL in normal populations as well as patients suffering illnesses and estimating the relative burden of different diseases. 11-13

All patients are expected to spend within 30 minutes on questionnaire survey.

In order to study for test-retest reliability, patient with endometriosis and adenomyosis scheduled for operation will be asked to complete the first set of questionnaires, EHP-30 and SF-36, when they attend for the pre-operative assessment clinic. The same set of EHP-30 will be completed when they are admitted for operation. In order to study the measurement properties of the questionnaire, the same set of EHP-30 and SF-36 will be given at the usual postoperative follow up visit which is usually scheduled 3-6 months later.

In order to study for test-retest reliability, patient with endometriosis and adenomyosis not scheduled for operation will be asked to complete the first set of questionnaires, EHP-30 and SF-36, at recruitment and a set of EHP-30 will be completed 2 weeks later and return by the return envelope provided. In order to study the measurement properties of the questionnaire, the same set of EHP-30 and SF-36 will be given at the usual gynaecology follow up visit which is usually scheduled 3-6 months after treatment.

All patients will be asked to report any important health or life changes that occur between the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Hong Kong Chinese women
* diagnosed with endometriosis or adenomyosis.

Exclusion Criteria:

* uterine fibroid more than 5 cm
* other premalignant or malignant conditions

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Eligible Chinese women attending the Gynaecology clinic of New Territories East Cluster will be invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Validation of Endometriosis health profile-30 (EHP-30) traditional Chinese (Hong Kong) version | Baseline
  internal consistency and construct validity

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ying Fung, Principal Investigator — 852-35052748
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided